CLINICAL TRIAL: NCT00005824
Title: Pilot Study of the Safety and Feasibility of Autologous Peripheral Blood Stem Cell Transplantation for Patients With Relapsed AIDS-Related Lymphoma
Brief Title: Chemotherapy Followed By Peripheral Stem Cell Transplantation in Treating Patients With Recurrent or Refractory AIDS-Related Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: AMC-020; CDR0000067835 (Other: NCI)
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Lymphoma
Keywords: AIDS-related peripheral/systemic lymphoma; AIDS-related diffuse large cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related small noncleaved cell lymphoma; HIV-associated Hodgkin lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related lymphoblastic lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Filgrastim; Busulfan; Cyclophosphamide; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: busulfan
Drug: cyclophosphamide
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy followed by peripheral stem cell transplantation in treating patients who have recurrent or refractory AIDS-related lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of intensive chemotherapy and autologous peripheral blood stem cell transplantation in patients with recurrent or refractory AIDS-related lymphoma.
* Determine the response and response duration in these patients treated with this regimen.
* Determine the effect of this treatment regimen on HIV RNA and CD4 cells in these patients.

OUTLINE: Patients receive mobilization chemotherapy consisting of cyclophosphamide IV over 2 hours followed 2 days later by daily filgrastim (G-CSF) subcutaneously (SC) until blood counts recover. Patients then undergo leukopheresis to collect CD34+ cells.

Patients receive conditioning chemotherapy consisting of oral busulfan every 6 hours on days -7, -6, -5, and -4 for a total of 14 doses and cyclophosphamide IV over 1 hour on days -3 and -2. Patients undergo autologous stem cell infusion on day 0. G-CSF is administered IV or SC daily beginning on day 1 and continuing until blood counts recover.

Patients are followed monthly for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 5-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Intermediate- or high-grade non-Hodgkin's lymphoma or Hodgkin's disease

  * Failed to achieve complete remission with initial therapy OR
  * Relapsed after initial therapy
* May be in complete remission after salvage therapy
* Sensitive to most recent chemotherapy

  * Improvement of at least 25% in bidimensional tumor measurements OR
  * Improvement in evaluable disease sustained over 4 weeks
* Measurable or evaluable disease
* HIV-1 positive
* CD4 greater than 50 cells/mm^3 (unless not receiving optimal antiretroviral therapy)
* HIV RNA less than 110,000 copies/mL (unless not receiving optimal antiretroviral therapy)
* No active leptomeningeal or parenchymal CNS involvement NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* Physiologic 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3

Hepatic:

* AST no greater than 3 times upper limit of normal
* Bilirubin no greater than 2.0 mg/dL (unless receiving indinavir)

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No history of cardiac disease
* LVEF at least 45%

Pulmonary:

* No history of symptomatic pulmonary disease
* DLCO at least 60%

Other:

* No active opportunistic infections
* No cytomegalovirus retinitis or pneumonitis requiring maintenance therapy
* No sensitivity to E. coli-derived products
* Not pregnant
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 1 week since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* Chronic suppressive therapy for infection allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-11; Primary Completion 2004-07 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David T. Scadden, MD, Study Chair — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts

REFERENCES:
- [Result] Spitzer TR, Ambinder RF, Lee JY, Kaplan LD, Wachsman W, Straus DJ, Aboulafia DM, Scadden DT. Dose-reduced busulfan, cyclophosphamide, and autologous stem cell transplantation for human immunodeficiency virus-associated lymphoma: AIDS Malignancy Consortium study 020. Biol Blood Marrow Transplant. 2008 Jan;14(1):59-66. doi: 10.1016/j.bbmt.2007.03.014. PMID 18158962